CLINICAL TRIAL: NCT01698970
Title: Effect of the Consumption of a Probiotic Strain on the Prevention of Post-operative Recurrence in Crohn's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: NU098
Record Dates: First submitted 2012-10-01; First posted 2012-10-03 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Crohn's Disease
Keywords: Probiotic; capsules; Crohn's disease; recurrent endoscopic ileo-colonic lesions
MeSH Terms: conditions — Crohn Disease | interventions — Capsules

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 = Tested product (Experimental)
  Interventions: Other: 1-Freeze-dried Probiotics provided in capsule (150 mg) containing 1,0x10E10 colony forming unit per capsule (test)
- 2 = Control product (Placebo Comparator)
  Interventions: Other: 2- excipients (150 mg) in capsule (control)

INTERVENTIONS:
Other: 1-Freeze-dried Probiotics provided in capsule (150 mg) containing 1,0x10E10 colony forming unit per capsule (test) — 1- 6 test products/day
  Arms: 1 = Tested product
Other: 2- excipients (150 mg) in capsule (control) — 2- 6 control poducts/day
  Arms: 2 = Control product

SUMMARY:
A double-blind, multicentre, stratified by centre, randomised, parallel study with two groups of adult patients operated on for Crohn's disease, to determine if oral ingestion of probiotics could prevent the appearance of Crohn's disease recurrent endoscopic ileo-colonic lesions 12 months after surgery. Patients will consume 900 mg/day of active product (N=56) or control product (N=56) during one year.

ELIGIBILITY:
Inclusion Criteria:

* Male/female at least 18 years old
* Diagnosis of Crohn's disease defined by the criteria usually adopted (Gower-Rousseau, 1994)
* Crohn's disease mainly limited to the terminal ileum and/or the ascending and transverse colon
* Diagnosis of Crohn's disease in agreement with surgical specimen analysis
* Patient having given its written consent to take part in the study
* Complete resection of all main macroscopic ileo-colonic lesions, as shown by inspection at surgery
* To have an ileo-colic resection (right, transverse, left) with an anastomosis that can be inspected by endoscopy
* Ability to start oral nutrition and therefore the consumption of the study product within 21 days of surgery
* Patient receiving no antibiotics at the beginning of the product consumption

Exclusion Criteria:

* One or more intestinal resection during the 5 last years before the last surgery
* Presence of any severe additional disease
* For female patient : pregnancy or breast feeding
* For pre-menopausal female patient : no effective contraceptive methods used (combined oestrogen-progestogen pill or Intrauterine Device)
* Patient currently in an exclusion period following participation in another clinical trial
* Patient in a situation which in the investigator's opinion could interfere with optimal participation in the present study or could constitute a special risk for the patient
* Significant presence of Crohn's disease in other intestinal tracts
* Small bowel cumulative resection exceeding 1 meter
* Patient with ileostomy
* Subtotal colectomy with ileo-rectal anastomosis
* Severe post-operative septic complications (fistula, peritonitis), leading to administration of more than 15 days of post-operative antibiotherapy)
* Intake of unauthorised treatments (mesalazine, olsalazine or sulfasalazine, 5-Aminosalicylates (5-ASA) or 4-Aminosalicylates (4-ASA)) ; corticoïds and immunosuppressors) after surgery except corticoids which will have to be stopped within 6 weeks after surgery according to standardised stepwise dose reductions
* Patient under artificial nutrition
* Subject with a loss of personal liberty, by administrative or judicial decision, or major with a legal guardian

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2004-02; Primary Completion 2007-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Huriez - Service des maladies de l'appareil digestif et de la nutrition, Lille, France